CLINICAL TRIAL: NCT05830799
Title: A Single-centre, Open-label, Fixed-sequence Trial to Evaluate the Impact of C21 on the Exposure of CYP1A2, CYP2C9, CYP3A4 and P-gp Substrates in Healthy Volunteers
Brief Title: A Trial to Evaluate the Impact of C21 on the Exposure of 4 Substrates in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VP-C21-012
Record Dates: First submitted 2023-03-24; First posted 2023-04-26 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Drug Interactions; Caffeine; Tolbutamide; Midazolam; nintedanib

STUDY DESIGN:
Intervention Model Description: Open label, one group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: C21 (Experimental): C21, single dose, oral administration twice daily, for 15 days
  Interventions: Drug: Drug Drug Interaction

INTERVENTIONS:
Drug: Drug Drug Interaction — The intervention phase consists of 3 periods: in period 1, the pharmacokinetics (PK) of all substrates will be evaluated in the absence of C21, in period 2, a potential inhibitory effect of C21 on the substrates be evaluated, and in period 3, the net effect of potential C21-mediated induction and inhibition on the substrates will be evaluated
  Other Names: Caffeine, Koffein Meda; Tolbutamide, Tolbutamide CF; Midazolam, Midazolam APL; Nintedanib, Ofev

SUMMARY:
This is a single-centre, open-label, fixed-sequence trial to evaluate the impact of C21 on the exposure of CYP1A2, CYP2C9, CYP3A4 and P-gp substrates in healthy volunteers.

DETAILED DESCRIPTION:
This is a single-centre, open-label, fixed-sequence trial to evaluate the influence of C21 on the exposure of CYP1A2, CYP2C9, CYP3A4 and P-gp substrates in healthy male and female volunteers.

The trial consists of a screening phase (Day -28 to Day -1), an open-label intervention phase (Day -1 to Day 19), and a follow-up phase (Day 20 to Day 25 [±2 days]). Subjects will remain at the trial site from the afternoon of Day -1 to the morning of Day 6, and again from the afternoon of Day 16 to the morning of Day 19.

The intervention phase consists of 3 periods: in period 1 (Day -1 to Day 3), the pharmacokinetics (PK) of all substrates will be evaluated in the absence of C21, in period 2 (Day 4 to Day 6), a potential inhibitory effect of C21 on the substrates be evaluated, and in period 3 (Day 17 to Day 19), the net effect of potential C21-mediated induction and inhibition on the substrates will be evaluated.

Subjects will be expected to attend a total of 4 visits to the trial site, including a screening visit (Visit 1), 2 intervention visits (Visits 2 and 3) and a follow-up visit (Visit 4).

Each subject is expected to participate in the trial for approximately 55 days, including an up to 28-day screening period, 19-day intervention period and a 4- to 8-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial.
2. Healthy male, or healthy female subject of non-childbearing potential, aged 18 to 60 years, inclusive.
3. Body mass index ≥ 18.5 and ≤ 30.0 kg/m2 at the time of the screening visit.
4. Medically healthy subject without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of the screening visit, as judged by the Investigator.
5. Women of non-childbearing potential, i.e. pre-menopausal females who have undergone any of the following surgical procedures; hysterectomy, bilateral salpingectomy or bilateral oophorectomy, or who are post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] >25 IU/L is confirmatory).
6. Male subjects who are vasectomised, who are willing to use condoms or to practice sexual abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the subject) to prevent pregnancy and drug exposure of a partner. Male subjects must also refrain from donating sperm from the first administration of IMP until 3 months after the last administration of IMP. Any female partner of a non-vasectomised male subject who is of child-bearing potential must use contraceptive methods with a failure rate of < 1% (see inclusion criterion no. 5) to prevent pregnancy from at least 2 weeks prior to the first administration of IMP to 4 weeks after the last administration of IMP.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the trial, or influence the results or the subject's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
3. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the trial.
5. Subjects who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
6. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
7. After 10 minutes supine rest at the screening visit, any vital signs values outside the following ranges:

   * Systolic blood pressure: <90 or >140 mmHg, or
   * Diastolic blood pressure <50 or >90 mmHg, or
   * Pulse <40 or >90 bpm
8. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the screening visit, as judged by the Investigator.
9. CYP2C9 genotype hetero- or homozygous for CYP2C9*2 (Arg144Cys) and/or CYP2C9*3 (Ile359Leu) variant alleles associated with altered CYP2C9 activity and tolbutamide metabolism [14], sampled at the screening visit.
10. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to any of the IMPs.
11. Regular use of any prescribed or non-prescribed medications, including antacids, analgesics, herbal remedies, e.g. St. John's wort, vitamins and minerals, within 2 weeks prior to the first administration of IMP, except occasional intake of paracetamol (maximum 2000 mg/day and not exceeding 3000 mg/week), as well as nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
12. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Subjects consented and screened but not dosed in previous phase 1 studies are not to be excluded.
13. Regular current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times/week is allowed before the screening visit.
14. Positive screening result for drugs of abuse or alcohol at the screening visit or on admission to the trial site prior to the first administration of the IMP.
15. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
16. Presence or history of drug abuse, as judged by the Investigator.
17. History of, or current use of anabolic steroids, as judged by the Investigator.
18. Excessive caffeine consumption defined by a daily intake of > 5 cups (1 cup = approximately 240 mL) of caffeine containing beverages, as judged by the Investigator.
19. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during the last three months prior to screening.
20. The Investigator considers the subject unlikely to comply with trial procedures, restrictions and requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Björn Schultze, MD, Principal Investigator — CTC Clinical Trial Consultants AB; Måns Jergil, PhD, Study Director — CTC Clinical Trial Consultants AB
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from CTC's database of volunteers and from strategic marketing campaigns (including social media).
Pre-assignment Details: In total, 36 prospective trial subjects were screened for inclusion. Of these, 14 subjects were screening failures (ineligible), 2 subjects withdrew consent, and 1 subject met the eligibility criteria but was not needed. Nineteen (19) subjects were included in the trial. Of the 19 included subjects, 18 subjects were fully evaluable, i.e., completed the trial up until at least the end of Day 19.
Period: Overall Study
Arm/Group | Experimental: C21
Started | 19
Completed | 18
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: C21
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 19

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Caffeine and Paraxanthine (Cmax)
Description: Maximum observed concentration (Cmax) for caffeine and its metabolite paraxanthine.
Time Frame: Pre-dose and 0:15, 0:30, 0:45, 1, 1:30, 2, 3, 4, 5, 6, 8, 12, 16, 24 hours post dose at Day 2 (period 1), Day 5 (period 2) and Day 18 (period 3)
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Period 1 - Without C21: In period 1 (Day 1 to Day 3), the pharmacokinetics (PK) of all substrates were evaluated in the absence of C21.
- Period 2 - With C21: In period 2 (Day 4 to Day 6), a potential inhibitory effect of C21 on the substrates was evaluated.
- Period 3 - With C21: In period 3 (Day 17 to Day 19), the net effect of potential C21-mediated induction and inhibition on the substrates was evaluated.
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
ng/mL
  Caffeine: number analyzed (Participants) | 18 | 18 | 17
  Caffeine | 2290 (22.3) | 2871 (18.7) | 2784 (37.1)
  Paraxanthine: number analyzed (Participants) | 18 | 18 | 17
  Paraxanthine | 546.4 (15.6) | 191.0 (43.5) | 467.7 (24.2)

2. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Caffeine and Paraxanthine (Tmax)
Description: Time of occurrence of Cmax (Tmax) for caffeine and its metabolite paraxanthine.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
hours
  Caffeine: number analyzed (Participants) | 18 | 18 | 17
  Caffeine | 0.6333 [0.500 to 1.00] | 0.7500 [0.250 to 2.00] | 0.5167 [0.250 to 4.00]
  Paraxanthine: number analyzed (Participants) | 18 | 18 | 17
  Paraxanthine | 6.000 [2.00 to 12.0] | 23.93 [12.0 to 24.0] | 11.90 [1.00 to 23.5]

3. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Caffeine and Paraxanthine (AUC0-last)
Description: Area under the plasma concentration vs. time curve from 0 to time of last measurable plasma concentration (AUC0-last) for caffeine and its metabolite paraxanthine.
Time Frame: Day 2 to day 19
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Caffeine: number analyzed (Participants) | 18 | 18 | 17
  Caffeine | 15760 (39.8) | 47560 (14.7) | 34690 (46.0)
  Paraxanthine: number analyzed (Participants) | 18 | 18 | 17
  Paraxanthine | 8667 (21.4) | 3013 (46.1) | 8285 (25.3)

4. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Caffeine and Paraxanthine (AUC0-inf)
Description: Area under the plasma concentration vs. time curve from 0 to infinity (AUC0-inf) for caffeine and its metabolite paraxanthine.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Caffeine: number analyzed (Participants) | 18 | 18 | 17
  Caffeine | 16880 (43.5) | 130500 (37.8) | 50190 (79.5)
  Paraxanthine: number analyzed (Participants) | 18 | 18 | 1
  Paraxanthine | 11020 (35.8) | NA (NA) — NA Explanation: Not calculated. Due to the shape of the paraxanthine plasma concentration vs. time curves in periods 2 and 3, Lambdaz could only be calculated for 2 subjects, hence summary statistics for the Lambdaz-dependent PK parameter AUC0-inf could not be calculated. | NA (NA) — NA Explanation: Not calculated. Due to the shape of the paraxanthine plasma concentration vs. time curves in periods 2 and 3, Lambdaz could only be calculated for 2 subjects, hence summary statistics for the Lambdaz-dependent PK parameter AUC0-inf could not be calculated.

5. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Tolbutamide and 4-hydroxy-tolbutamide and Carboxy-tolbutamide (Cmax)
Description: Maximum observed concentration (Cmax) for Tolbutamide and its metabolites 4-hydroxy-tolbutamide and carboxy-tolbutamide.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
ng/mL
  Tolbutamide | 48390 (9.75) | 61070 (15.2) | 64130 (15.4)
  4-Hydroxy-Tolbutamide | 670.5 (27.8) | 25.49 (83.0) | 88.71 (63.5)
  Carboxy-Tolbutamide | 2040 (25.2) | 81.35 (96.2) | 256.3 (76.4)

6. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Tolbutamide and 4-hydroxy-tolbutamide and Carboxy-tolbutamide (Tmax)
Description: Time of occurrence of Cmax (Tmax) for Tolbutamide and its metabolites 4-hydroxy-tolbutamide and carboxy-tolbutamide.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
hours
  Tolbutamide | 2.500 [1.50 to 4.10] | 4.000 [2.00 to 24.0] | 4.000 [1.50 to 8.02]
  4-Hydroxy-Tolbutamide | 4.000 [2.00 to 8.02] | 15.23 [8.00 to 24.0] | 11.91 [8.00 to 23.7]
  Carboxy-Tolbutamide | 4.000 [2.00 to 6.00] | 11.98 [8.00 to 24.0] | 11.90 [8.00 to 23.7]

7. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Tolbutamide and 4-hydroxy-tolbutamide and Carboxy-tolbutamide (AUC0-last)
Description: Area under the plasma concentration vs. time curve from 0 to time of last measurable plasma concentration (AUC0-last) for Tolbutamide and its metabolites 4-hydroxy-tolbutamide and carboxy-tolbutamide.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Tolbutamide | 449800 (15.8) | 1146000 (16.3) | 1207000 (18.8)
  4-Hydroxy-Tolbutamide | 6872 (23.6) | 316.8 (51.6) | 960.5 (47.7)
  Carboxy-Tolbutamide | 21800 (20.7) | 1034 (62.3) | 2729 (59.3)

8. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Tolbutamide and 4-hydroxy-tolbutamide and Carboxy-tolbutamide (AUC0-inf)
Description: Area under the plasma concentration vs. time curve from 0 to infinity (AUC0-inf) for Tolbutamide and its metabolites 4-hydroxy-tolbutamide and carboxy-tolbutamide.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Tolbutamide: number analyzed (Participants) | 18 | 17 | 18
  Tolbutamide | 499100 (19.3) | 9919000 (71.2) | 6134000 (69.2)
  4-Hydroxy-Tolbutamide | 8142 (24.1) | NA (NA) — Not calculated. Due to the shape of the 4-hydroxy-tolbutamide and carboxy-tolbutamide plasma concentration vs. time curves in periods 2 and 3, Lambdaz could not be calculated and subsequently, summary statistics for the Lambdaz-dependent PK parameter AUC0-inf for the tolbutamide metabolites in these trial periods could not be calculated. | NA (NA) — Not calculated. Due to the shape of the 4-hydroxy-tolbutamide and carboxy-tolbutamide plasma concentration vs. time curves in periods 2 and 3, Lambdaz could not be calculated and subsequently, summary statistics for the Lambdaz-dependent PK parameter AUC0-inf for the tolbutamide metabolites in these trial periods could not be calculated.
  Carboxy-Tolbutamide | 24790 (18.0) | NA (NA) — Not calculated. Due to the shape of the 4-hydroxy-tolbutamide and carboxy-tolbutamide plasma concentration vs. time curves in periods 2 and 3, Lambdaz could not be calculated and subsequently, summary statistics for the Lambdaz-dependent PK parameter AUC0-inf for the tolbutamide metabolites in these trial periods could not be calculated. | NA (NA) — Not calculated. Due to the shape of the 4-hydroxy-tolbutamide and carboxy-tolbutamide plasma concentration vs. time curves in periods 2 and 3, Lambdaz could not be calculated and subsequently, summary statistics for the Lambdaz-dependent PK parameter AUC0-inf for the tolbutamide metabolites in these trial periods could not be calculated.

9. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Midazolam and 1-hydroxy-midazolam (Cmax)
Description: Maximum observed concentration (Cmax) for midazolam and its metabolite 1-hydroxy-midazolam.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
ng/mL
  Midazolam | 10.89 (33.1) | 14.32 (36.4) | 12.69 (25.8)
  1-Hydroxy-Midazolam | 3.187 (50.2) | 3.175 (52.5) | 2.570 (50.9)

10. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Midazolam and 1-hydroxy-midazolam (Tmax)
Description: Time of occurrence of Cmax (Tmax) for midazolam and its metabolite 1-hydroxy-midazolam.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
hours
  Midazolam | 0.7500 [0.500 to 0.783] | 0.7500 [0.500 to 1.00] | 0.7500 [0.500 to 1.00]
  1-Hydroxy-Midazolam | 0.7500 [0.500 to 1.00] | 0.7500 [0.500 to 1.50] | 0.7500 [0.500 to 1.00]

11. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Midazolam and 1-hydroxy-midazolam (AUC0-last)
Description: Area under the plasma concentration vs. time curve from 0 to time of last measurable plasma concentration (AUC0-last) for midazolam and its metabolite 1-hydroxy-midazolam.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Midazolam | 29.17 (39.6) | 42.06 (35.4) | 35.09 (28.9)
  1-Hydroxy-Midazolam | 7.835 (41.9) | 8.695 (39.6) | 6.465 (41.4)

12. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Midazolam and 1-hydroxy-midazolam (AUC0-inf)
Description: Area under the plasma concentration vs. time curve from 0 to to infinity (AUC0-inf) for midazolam and its metabolite 1-hydroxy-midazolam.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Midazolam | 30.41 (39.7) | 43.77 (35.8) | 36.58 (28.9)
  1-Hydroxy-Midazolam | 8.700 (39.7) | 9.756 (39.3) | 7.316 (40.2)

13. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Nintedanib and BIBF 1202 (Cmax)
Description: Maximum observed concentration (Cmax) for nintedanib and its metabolite BIBF 1202.
Time Frame: Pre-dose and 0:15, 0:30, 0:45, 1, 1:30, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48 hours post dose at Day 1 (period 1), Day 4 (period 2) and Day 17 (period 3)
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
ng/mL
  Nintedanib: number analyzed (Participants) | 18 | 18 | 17
  Nintedanib | 10.10 (80.4) | 13.87 (79.0) | 13.72 (61.3)
  BIBF 1202: number analyzed (Participants) | 18 | 18 | 17
  BIBF 1202 | 12.03 (97.7) | 15.16 (66.7) | 13.61 (90.8)

14. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Nintedanib and BIBF 1202 (Tmax)
Description: Time of occurrence of Cmax (Tmax) for nintedanib and its metabolite BIBF 1202.
Time Frame: as for outcome 13
Population: PK analysis set.
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
hours
  Nintedanib: number analyzed (Participants) | 18 | 18 | 17
  Nintedanib | 3.000 [1.00 to 6.07] | 3.000 [1.00 to 6.00] | 2.000 [0.767 to 6.00]
  BIBF 1202: number analyzed (Participants) | 18 | 18 | 17
  BIBF 1202 | 4.000 [2.00 to 6.02] | 4.000 [1.52 to 6.00] | 3.033 [2.00 to 6.00]

15. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Nintedanib and BIBF 1202 (AUC0-last)
Description: Area under the plasma concentration vs. time curve from 0 to time of last measurable plasma concentration (AUC0-last) for nintedanib and its metabolite BIBF 1202.
Time Frame: as for outcome 13
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Nintedanib: number analyzed (Participants) | 18 | 18 | 17
  Nintedanib | 92.87 (82.3) | 128.4 (57.9) | 106.4 (48.2)
  BIBF 1202: number analyzed (Participants) | 18 | 18 | 17
  BIBF 1202 | 103.1 (102) | 133.1 (59.1) | 106.8 (68.8)

16. Primary Outcome: To Evaluate the Impact of C21 on the Pharmacokinetics (PK) of Nintedanib and BIBF 1202 (AUC0-inf)
Description: Area under the plasma concentration vs. time curve from 0 to infinity (AUC0-inf) for nintedanib and its metabolite BIBF 1202.
Time Frame: as for outcome 13
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 18 | 18 | 18
h*ng/mL
  Nintedanib: number analyzed (Participants) | 18 | 18 | 17
  Nintedanib | 101.0 (80.3) | 143.3 (56.2) | 114.7 (47.4)
  BIBF 1202: number analyzed (Participants) | 18 | 18 | 17
  BIBF 1202 | 110.1 (98.9) | 141.8 (58.9) | 113.8 (63.6)

17. Secondary Outcome: To Evaluate the Pharmacokinetics (PK) of C21 and M1 (Cmax)
Description: Maximum observed concentration (Cmax) of C21 and its main metabolite M1.
Time Frame: Day 17
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Experimental: C21
Number analyzed (Participants) | 18
ng/mL
  C21: number analyzed (Participants) | 17
  C21 | 1433 (55.7)
  M1: number analyzed (Participants) | 17
  M1 | 421.6 (29.1)

18. Secondary Outcome: To Evaluate the Pharmacokinetics (PK) of C21 and M1 (Tmax)
Description: Time of occurrence of Cmax (Tmax) of C21 and its main metabolite M1.
Time Frame: Day 17
Population: PK analysis set.
Measure: Median (Full Range); unit: hours
Arm/Group | Experimental: C21
Number analyzed (Participants) | 18
hours
  C21: number analyzed (Participants) | 17
  C21 | 1.000 [0.500 to 2.00]
  M1: number analyzed (Participants) | 17
  M1 | 3.000 [2.00 to 4.00]

19. Secondary Outcome: To Evaluate the Pharmacokinetics (PK) of C21 and M1 (AUC0-last)
Description: Area under the plasma concentration vs. time curve from 0 to time of last measurable plasma concentration (AUC0-last) of C21 and its main metabolite M1.
Time Frame: Day 17
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Experimental: C21
Number analyzed (Participants) | 18
h*ng/mL
  C21: number analyzed (Participants) | 17
  C21 | 2041 (30.4)
  M1: number analyzed (Participants) | 17
  M1 | 2731 (37.6)

20. Secondary Outcome: To Evaluate the Pharmacokinetics (PK) of C21 and M1 (AUC0-tau)
Description: Area under the plasma concentration vs. time curve from 0 to the end of the dosing interval (AUC0-tau) of C21 and its main metabolite M1.
Time Frame: Day 17
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Experimental: C21
Number analyzed (Participants) | 18
h*ng/mL
  C21: number analyzed (Participants) | 17
  C21 | 2049 (30.3)
  M1: number analyzed (Participants) | 17
  M1 | 2734 (37.5)

21. Secondary Outcome: To Evaluate the Safety of C21 (AEs)
Description: Frequency, seriousness and intensity of adverse events (AEs).
Time Frame: From signing ICF to Day 25
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
Number analyzed (Participants) | 19 | 18 | 18
Participants
  Any AE | 8 | 10 | 5
  Any SAE | 0 | 0 | 0
  Any AE leading to withdrawal from trial | 0 | 0 | 0
  Any AE leading to death | 0 | 0 | 0
  Causality - C21 - Related | 0 | 7 | 3
  Causality - C21 - Not Related | 1 | 5 | 13
  Causality - C21 - Not Applicable | 7 | 0 | 2
  Causality - Nintedanib - Related | 4 | 5 | 2
  Causality - Nintedanib - Not Related | 4 | 7 | 2
  Causality - Nintedanib - Not Applicable | 0 | 2 | 1
  Causality - Caffeine - Related | 1 | 5 | 0
  Causality - Caffeine - Not Related | 3 | 8 | 3
  Causality - Caffeine - Not Applicable | 4 | 2 | 3
  Causality - Tolbutamide - Related | 1 | 5 | 0
  Causality - Tolbutamide - Not Related | 3 | 8 | 4
  Causality - Tolbutamide - Not Applicable | 4 | 2 | 3
  Causality - Midazolam - Related | 1 | 5 | 0
  Causality - Midazolam - Not Related | 3 | 8 | 4
  Causality - Midazolam - Not Applicable | 4 | 2 | 3
  Severity - Mild | 7 | 9 | 4
  Severity - Moderate | 1 | 3 | 1
  Severity - Severe | 0 | 0 | 0
  Severity - Life-Threatening | 0 | 0 | 0
  Severity - Death | 0 | 0 | 0

22. Secondary Outcome: To Evaluate the Safety of C21 (Vital Signs)
Description: Number of patients with clinically significant changes in vital signs (systolic and diastolic blood pressure and pulse) from baseline. Any vital signs outside of normal ranges were judged as clinically significant or not clinically significant
Time Frame: From screening to day 25
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: C21
Number analyzed (Participants) | 19
Participants | 0

23. Secondary Outcome: To Evaluate the Safety of C21 (ECG)
Description: Number of patients with clinically significant changes in electrocardiogram (ECG) from baseline. The resting heart rate (HR) and PQ/PR, QRS, QT and QTcF intervals were recorded. Any abnormalities were specified and documented as clinically significant or not clinically significant
Time Frame: From screening to day 25
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: C21
Number analyzed (Participants) | 19
Participants | 0

24. Secondary Outcome: To Evaluate the Safety of C21 (Clinical Laboratory Measurements)
Description: Number of patients with clinically significant changes in clinical laboratory measurements (haematology, clinical chemistry, coagulation) from baseline. Any laboratory values outside of normal ranges were specified and documented as normal, abnormal not clinically significant, or abnormal clinically significant.
Time Frame: From screening to day 25
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: C21
Number analyzed (Participants) | 19
Participants | 0

ADVERSE EVENTS:
Time Frame: From signing ICF to Day 25
Arm/Group | Period 1 - Without C21 | Period 2 - With C21 | Period 3 - With C21
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 8/19 | 10/18 | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1 - Without C21 (N=19) | Period 2 - With C21 (N=18) | Period 3 - With C21 (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 5 (8) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT05830799/Prot_SAP_000.pdf